CLINICAL TRIAL: NCT01022801
Title: A Phase II Study in Japan of the Safety and Antiviral Activity of Entecavir (BMS-200475) vs Lamivudine in Adults With Chronic Hepatitis B Infection
Brief Title: A Phase II Dose Response Study in Japan in Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI463-047
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Entecavir (0.01 mg) (Experimental)
  Interventions: Drug: Entecavir
- Entecavir (0.1 mg) (Experimental)
  Interventions: Drug: Entecavir
- Entecavir (0.5 mg) (Experimental)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Capsule, P.O., 0.01, 0.1 or 0.5 mg, once daily for 24 weeks
  Other Names: Baraclude; BMS-200475

SUMMARY:
To demonstrate the dose response of entecavir in Japanese patients as measured by HBV DNA levels by PCR (log10 copies/mL) at Week 22

ELIGIBILITY:
Inclusion Criteria:

* Positive for HBsAg OR, negative for IgM core antibody and confirmation of chronic hepatitis B on liver biopsy,
* Positive for HBeAg OR negative for HBeAg with positive HBeAb,
* Documented HBV Viremia on 2 or more occasions: Viremia on sample drawn AND HBV DNA of ≥ 40 MEq/mL by Quantiplex assay at the screening visit

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-08; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in HBV DNA levels as measured by by PCR (log10 copies/mL) | at Week 22

SECONDARY OUTCOMES:
Incidence of clinical adverse events and discontinuations due to adverse events in each entecavir group in comparison to lamivudine | Through Week 24 (end of dosing) plus 5 days
Incidence of laboratory abnormalities in each entecavir group in comparison to lamivudine | Through Week 24 (end of dosing) plus 5 days
HBV DNA as measured by PCR (log10 copies/mL) at Week 22 [to demonstrate non-inferiority of at least one dose of entecavir as compared with lamivudine] | Week 22
Proportion of subjects in each treatment group who achieve HBV DNA reduced by ≥2 log10 and/or below the limit of quantification (LOQ) (<400 copies/mL) as measured by PCR assay | Week 12, Week 22
Proportion of subjects in each treatment group who achieve HBV DNA below the limit of detection (0.7 MEq/mL) of the Quantiplex branched DNA hybridization assay (Quantiplex assay) | Week 22
Proportion of subjects in each treatment group who achieve normalization of ALT (ALT <1.25 x UKN) | Week 22
Proportion of subjects in each treatment group who achieve loss of HBeAg at Week 22 among HBeAg-positive subjects at baseline | Baseline, Week 22
Proportion of subjects in each treatment group who achieve seroconversion at Week 22 among of HBeAg-positive subjects at baseline | Week 22
Proportion of HBeAg-positive subjects at baseline who achieve responder status (defined as: HBV DNA <0.7 MEq/mL by the Quantiplex assay; loss of HBeAg and normal serum ALT) | Week 22
Proportion of HBeAg-negative subjects at baseline who achieve responder status (defined as HBV DNA <0.7 MEq/mL by the Quantiplex assay and normal serum ALT) | Week 22
Incidence of genotypic resistance of HBV isolates in subjects who have a ε 1 log10 increase in HBV DNA as measured by PCR assay after achieving the lowest value while on study drug | Through Week 24
Relationship of HBV isolates (genotypes A, B, C etc) at baseline compared to response | Week 22

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx